CLINICAL TRIAL: NCT05317494
Title: A Prospective Non-Interventional Study to Describe the Effectiveness and Safety of Venetoclax as a First-Line Treatment in Acute Myeloid Leukemia (AML) Patients Who Are Ineligible to Intensive Chemotherapy in Routine Clinical Practice in Greece
Brief Title: A Study to Assess Change in Disease State in Adult Participants With Acute Myeloid Leukemia (AML) Ineligible for Intensive Chemotherapy Receiving Oral Venetoclax Tablets in Greece
Acronym: SURVIVE
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P22-535
Record Dates: First submitted 2022-03-21; First posted 2022-04-07 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Venetoclax; Venclexta; Venclyxto; ABT-199; Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Venetoclax Participants: Participants treated with Venetoclax in accordance with approved local label.

SUMMARY:
Acute Myeloid Leukemia (AML) is a cancer of the blood and bone marrow and is the most common acute leukemia in adults. This study will evaluate how well Venetoclax works to treat AML in adult participants who are ineligible for intensive chemotherapy in Greece.

Venetoclax is a drug approved to treat Acute Myeloid Leukemia. All study participants will receive Venetoclax as prescribed by their study doctor in accordance with approved local label. Adult participants with a new diagnosis of AML who are ineligible for intensive chemotherapy will be enrolled.

Around 100 participants will be enrolled in the study in approximately 15 sites in Greece.

Participants will receive venetoclax tablets to be taken by mouth daily according to the approved local label. The duration of the study is approximately 30 months.

There is expected to be no additional burden for participants in this trial. All study visits will occur during routine clinical practice and participants will be followed for 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant diagnosed Acute Myeloid Leukemia (AML) who is ineligible to intensive chemotherapy and is eligible to receive venetoclax as a first-line therapy, as per Greek Ministry of Health (MOH) label.
* Physician has decided to initiate venetoclax treatment. The decision to treat with venetoclax is made by the physician in accordance with the local label prior to any decision to approach the patient to participate in this study.

Exclusion Criteria:

- Participating in an interventional clinical trial within 30 days prior to venetoclax treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with acute myeloid leukemia (AML) treated with venetoclax per approved local label in Greece.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Overall Survival (OS) | Up to 30 Months
  OS is defined as the time from treatment initiation to death from any cause.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Composite Complete Remission | Up to 30 Months
  Composite complete remission is defined as the proportion of participants with complete remission (CR) or complete remission with incomplete marrow recovery (CRi).
Total Time of Treatment with Venetoclax Combination Therapy | Up to 30 Months
  The total time of treatment with venetoclax combination therapy.
Time to Transfusion Independence | Up to 30 Months
  Total duration of transfusion independence is defined as the period of at least 56 days with no Red Blood Cell (RBC) or platelet transfusion between the first dose of study drug and the last dose of study drug plus 30 days.
Post Baseline RBC and Platelet Transfusion Independence Rate | Up to 30 Months
  Post baseline RBC and platelet transfusion independence rate will be calculated as the proportion of participants who achieved RBC and platelet, respectively, transfusion independence post baseline.
Change from Baseline in European Quality of Life 5 Dimensions (EQ-5D-5L) Considered Minimally Clinical Important | Up to 30 Months
  The EQ-5D-5L is a standardized instrument used to measure health-related quality of life that can be used in a wide range of health conditions and treatments.
Treatment Patterns Venetoclax in Combination with Hypomethylating Agents (HMAs) | Up to 30 Months
  Treatment patterns defined by the proportion of participants treated with venetoclax in combination with HMAs (dosing with venetoclax and any modifications/interruptions/titrations, type and dosing of each HMA, frequency of response assessment, cycle length, dosing, concomitant medications, etc).
Healthcare Resource Utilization as the Number of Transfusions (Red Blood Cell [RBC] or Platelets) Received during First-line Treatment in an Outpatient Setting | Up to 30 Months
  Healthcare resource utilization as the number of transfusions (red blood cell [RBC] or platelets) received during first-line treatment in an outpatient setting.
Healthcare Resource Utilization as the Number of Hospitalizations during First-line Treatment | Up to 30 Months
  Healthcare resource utilization as the number of hospitalizations during first-line treatment.
Healthcare Resource Utilization as the Number of Intensive Care Unit (ICU) Admissions during First-line Treatment | Up to 30 Months
  Healthcare resource utilization as the number of intensive care unit (ICU) admissions during first-line treatment.
Healthcare Resource Utilization as the Number of Visits in a Private Healthcare Practitioner | Up to 30 Months
  Healthcare resource utilization as the number of visits in a private healthcare practitioner.
Healthcare Resource Utilization as the Name of Relevant Medication due to Infections (Antibiotics or Other) | Up to 30 Months
  Healthcare resource utilization as the name of relevant medication due to infections (antibiotics or other).
Healthcare Resource Utilization as the Dosing Scheme of Relevant Medication due to Infections (Antibiotics or Other) | Up to 30 Months
  Healthcare resource utilization as the dosing scheme of relevant medication due to infections (antibiotics or other).
Healthcare Resource Utilization as the Number of Laboratory Tests | Up to 30 Months
  Healthcare resource utilization as the number of laboratory tests.
Healthcare Resource Utilization as the Type of Laboratory Tests | Up to 30 Months
  Healthcare resource utilization as the type of laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- Greece (13):
  - Olympion General Clinic /ID# 268392, Pátrai, Achaia
  - General Hospital of Athens Gennimatas /ID# 245968, Athens, Attica
  - General Hospital of Athens Laiko /ID# 244338, Athens, Attica
  - University General Hospital Attikon /ID# 248265, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 244337, Heraklion, Crete
  - General University Hospital of Alexandroupolis /ID# 244235, Alexandroupoli
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 244339, Athens
  - General Anti-cancer Hospital Agios Savvas /ID# 244408, Athens
  - General Hospital of Athens Laiko - Hematology Location /ID# 244234, Athens
  - University General Hospital of Ioannina /ID# 244336, Ioannina
  - University General Hospital of Patras /ID# 244335, RION Patras Achaia
  - Papageorgiou General Hospital /ID# 248266, Thessaloniki
  - General Hospital of Thessaloniki George Papanikolaou /ID# 244237, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info. — https://www.rxabbvie.com/